CLINICAL TRIAL: NCT06397703
Title: A Phase II Prospective 2-Arm Cohort Interventional Trial Utilizing Ultra-Hypofractionated SBRT With or Without Short Course Androgen Deprivation Therapy For Unfavorable Intermediate Risk Prostate Cancer
Brief Title: ADT and SBRT vs SBRT Alone for Unfavorable Intermediate Risk Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-01267
Record Dates: First submitted 2024-04-29; First posted 2024-05-03 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; relugolix; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ADT with SBRT (Experimental): The ADT patients will be treated with monthly Degarelix, or Leuprolide injections or daily Relugolix pills. After three months have elapsed, these patients as per routine will undergo SBRT. SBRT comprises stereotactic, ultra-fractionated radiotherapy every other day for five total treatments.
  Interventions: Drug: Leuprolide, Degarelix or Relugolix; Radiation: Stereotactic body radiation therapy/radiosurgery (SBRT)
- SBRT Alone (Active Comparator): Participants treated with SBRT alone (standard of care) will be administered stereotactic, ultra-fractionated radiotherapy every other day for five total treatments.
  Interventions: Radiation: Stereotactic body radiation therapy/radiosurgery (SBRT)

INTERVENTIONS:
Drug: Leuprolide, Degarelix or Relugolix — Patients assigned to the androgen deprivation therapy (ADT) arm will be treated with monthly Degarelix, or Leuprolide injections or daily Relugolix pills which are all standard ADT interventions.
  Arms: ADT with SBRT
Radiation: Stereotactic body radiation therapy/radiosurgery (SBRT) — SBRT will be directed to the prostate and delivered with a prescription dose of 40 Gy in 5 fractions prescribed to the 95% isodose line encompassing the planning target volume. Intra-fraction motion targeting and target position corrections will be utilized for each of the 5 treatment fractions.

SUMMARY:
For this study, unfavorable intermediate risk prostate cancer patients will select whether they are to be treated with the standard of care (SOC) 6 months of Androgen Deprivation Therapy (ADT) in conjunction with stereotactic body radiation therapy/radiosurgery (SBRT) directed to the prostate versus SBRT alone. The patient population will include those with National Comprehensive Cancer Network (NCCN)-defined unfavorable intermediate risk disease. All patients will be followed every 6 months for up to 5 years from the first patient treated and will undergo a routine 24-30 months post-SBRT prostate biopsy to assess for local tumor control.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven unfavorable intermediate risk prostate cancer, which includes patients with any one of the following variables: Gleason 4+3 disease; Percent positive cores > 50% of Gleason 7 disease; 2-3 intermediate risk factors (Gleason 7; PSA 10-20 ng/mL; or T2b-T2c)
* Patients must have tissue available for Decipher score testing. Results must be available before start of treatment.
* Serum testosterone ≥ 150 ng/dL determined within 2 months prior to enrollment
* At least 4 weeks must have elapsed from major surgery
* Karnofsky Performance Scale (KPS) ≥ 80%
* Prostate size as determined on MRI to be < 90 cc. Prostate size can be determined on CT scan if MRI is not available
* IPSS ≤ 20
* Patient must be available for follow-up. After 2 years of follow-up, upon completion of post-treatment biopsy, telephone and chart review-based follow-up will be acceptable
* Adequate hepatic function with serum bilirubin less than or equal to 1.5 times the upper institutional limits of normal (ULN), Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) less than or equal to 2.5 x ULN. Patients with a history of Gilbert's syndrome may be enrolled if the total bilirubin is < 3 mg/dL with a predominance of indirect bilirubin
* Adequate renal function with serum creatinine less than or equal to 1.5 x ULN
* Adequate hematologic function with absolute neutrophil counts of at least 1,500 cell/mm3 and platelets of at least 100,000 cells/mm3 and hemoglobin value > 9 g/dL (Note: patients whose anemia has been corrected to a hemoglobin value > 9 g/dL with blood transfusions are allowed).

Exclusion Criteria:

* CT or MRI or Positron Emission Tomography (PET) scan evidence of metastatic disease to the bone
* Patients with one or more positive lymph nodes considered suspicious as determined by clinical assessment on MRI or CT or PET scan
* Prior treatment for prostate cancer, including history of chemotherapy, hormonal therapy within 30 days of enrollment or surgery for prostate cancer (except for prior (transurethral resection of prostate) TURP or greenlight (photoselective vaporization of prostate) PVP which would be allowed)
* History of another malignancy within the previous 2 years except for the following: adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, currently in complete remission, or any other cancer that has been in complete remission for at least 3 years
* Patients with Crohn's disease or ulcerative colitis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2030-04-16 (Estimated); Study Completion 2031-04-16 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival | Up to Year 5
  Defined as the percentage of participants who survive without any signs or symptoms of prostate cancer.

SECONDARY OUTCOMES:
Incidence of Biochemical Failure | Up to Year 5
  Biochemical failure recurrence will be determined according to the established Phoenix criteria of 2 ng/nl elevation of the prostate specific antigen (PSA) nadir level (nadir + 2 definition).
Incidence of Distant Metastases | Up to Year 5
  Number of distant metastases observed over the course of the study.
Overall Survival | Up to Year 5
  Defined as the length of time from the date of first treatment until death.
Number of Positive Post-Treatment Biopsies | Year 2 Post-Treatment (Month 24-30)
Change in Expanded Prostate Cancer Index Composite (EPIC) Questionnaire Score (EPIC-26) | Baseline, Year 2
  26-item assessment of prostate cancer symptoms. Late bowel function as reported by the patient using the standardized questionnaire Expanded Prostate Cancer Index Composite (EPIC) sub-domain approximately 1 year after the end of treatment. The EPIC questionnaire contains 26 questions measuring patient function. Each question has a response option ranging from 0 or 1 (best) to 3, 4, or 5 (worst). The responses then correlate to a scoring scale of 0 to 100, where 0 is the best and 100 is the worst. The values vary from 0 to 100 for each question. The scores are averaged to derive a quality of life score, ranging from 0-100.
Change in International Prostatism Symptom Score (IPSS) | Baseline, Year 2
  7-item questionnaire of benign prostatic hyperplasia (BPH) symptoms. Each item is rated on a scale from 0 (not at all) to 5 (almost always). The total score is the sum of responses and ranges from 0 to 35; higher scores indicate greater BPH symptomology.
Change in 12-Item Short Form Health Survey (SF-12) Score | Baseline, Year 2
  The SF-12 is a 12-item assessment of the impact of health on an individual's everyday life. The total score is the sum of each item and is standardized; the total score ranges from 0 to 100, with higher scores indicated better physical and mental health functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zelefsky, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
De-identified IPD access will be limited to study team members who are IRB approved and listed on the delegation log.